CLINICAL TRIAL: NCT01954238
Title: A Phase I, Randomized, Double-blind, Placebo-controlled, Single and Multiple Sequential Ascending Dose Study Evaluating the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Orally Administered GCC-4401C in Healthy Males
Brief Title: A Study to Access Safety, Tolerability, Pharmacokinetics(PK) and Pharmacodynamics(PD) of Orally Administered GCC-4401C in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Green Cross Corporation (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Organization: GC Biopharma Corp (Industry)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: GC2107_102
Record Dates: First submitted 2013-09-23; First posted 2013-10-01 (Estimated); Last update posted 2014-12-23 (Estimated); Status verified 2014-12

CONDITIONS: Healthy Volunteers
Keywords: Anti-coagulant; Coagulation factor Xa inhibitor
MeSH Terms: interventions — Rivaroxaban

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Rivaroxaban (Active Comparator): Orally active direct factor Xa inhibitor for use in the prevention and treatment of venous thromboembolic disease
  Interventions: Drug: GCC-4401C
- Placebo (Placebo Comparator): GCC-4401C matching placebo capsule
  Interventions: Drug: GCC-4401C
- GCC-4401C (Experimental): Orally active direct factor Xa inhibitor for use in the prevention and treatment of venous thromboembolic disease. It is a novel molecule with a structural similarity to Rivaroxaban.
  Interventions: Drug: Rivaroxaban; Drug: Placebo

INTERVENTIONS:
Drug: GCC-4401C — * Orally active direct factor Xa inhibitor for use in the prevention and treatment of venous thromboembolic disease.
  * The dose selection for this clinical study was based on the safety, Pharmacokinetics and Pharmacodynamics results of the single dose study.
  * GCC-4401C was well tolerated in the single ascending dose study up to the highest single oral dose administered of 80 mg from 2.5 mg in 48 subjects.
  * The study consists of five cohorts (10 mg, 20 mg, 40 mg, 60 mg, and 80 mg) with eight subjects per cohort.
  * In the 20 mg cohort, six additional subjects will receive rivaroxaban (Xarelto®) 20 mg as an active comparator in open-label fashion.
  Other Names: Nokxaban
  Arms: Placebo; Rivaroxaban
Drug: Rivaroxaban — Rivaroxaban (Xarelto®) 20 mg tablets for oral administration IMP, placebo and comparator will be administered the same time points. The comparator will be administered open-label 30 minutes after a standard breakfast.
  Other Names: Xarelto
  Arms: GCC-4401C
Drug: Placebo — GCC-4401C matching placebo(Capsule): Strength is not applicable. GCC-4401C and placebo will be administered double-blind after a 10 hours fast.
  Other Names: GCC-4401C matching placebo
  Arms: GCC-4401C

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability and Pharmacokinetics/Pharmacodynamics of multiple doses of GCC-4401C in healthy male subjects.

DETAILED DESCRIPTION:
The primary objective is to investigate the safety, tolerability, and pharmacokinetics of multiple doses of GCC-4401C in healthy male subjects.

Forty-six subjects are planned for enrollment. The study consists of five cohorts (10 mg, 20 mg, 40 mg, 60 mg, and 80 mg) with eight subjects per cohort. In the 20 mg cohort, six additional subjects will receive rivaroxaban (Xarelto®) 20 mg as an active comparator in open-label fashion. Within each of the five cohorts, six subjects will be randomized to GCC-4401C and two subjects will be randomized to placebo.

The secondary objectives of this study are

* To characterize the single dose safety, tolerability, and PK after oral administration of GCC-4401C in healthy male subjects.
* To characterize the multiple dose pharmacodynamics after oral administration of GCC-4401C in healthy male subjects.
* To determine an appropriate dose range and dosing regimen of oral GCC-4401C for subsequent clinical trials.
* To compare the PK and PD of GCC-4401C with an active rivaroxaban (Xarelto®)group at 20 mg in healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Subject voluntarily has agreed to participate in this study and signed an Institutional Review Board (IRB)-approved informed consent before any of the Screening procedures will be performed.
2. Males between 18 to 45 years of age, inclusive, at Screening.
3. Non-smokers (or other nicotine use) as determined by history (no nicotine use over the past month prior to screening) and by urine cotinine concentration (< 400 ng/mL) at Screening.
4. Body mass index (BMI) between 18.5 and 28.0 kg/m2 at Screening.
5. Healthy, determined by pre-study medical evaluation and Investigator/designee discretion (medical history, physical examination, vital signs, ECG, and clinical laboratory evaluations).

Exclusion Criteria:

1. Clinically significant history or evidence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, neurological, immunological, or psychiatric disorder(s) as determined by the Investigator/designee.
2. Any disorder that would interfere with the absorption, distribution, metabolism, or excretion of drugs.
3. Have any of the following, which may put them at increased risk with anticoagulant use: family history or personal history of bleeding disorders or diseases/syndromes that can either alter or increase the propensity for bleeding; any other contraindication to anticoagulant treatment, or increased bleeding risk, as judged by the Investigator.
4. Are considering or scheduled to undergo any surgical procedure during the study.
5. Any concurrent disease or condition that, in the opinion of the Investigator/designee, would make the subject unsuitable for participation in the clinical study.
6. Fecal occult blood positive test at screening and admission.
7. Subject has history of alcohol and/or illicit drug abuse within one year of the Screening visit.
8. Positive Screening test for Hepatitis B surface antigen (HBsAg), Hepatitis C antibody, or human immunodeficiency virus (HIV) antibody.
9. Positive alcohol breathalyzer test at Screening or Day -1.
10. Positive urine drug test (cocaine, amphetamines, barbiturates, opiates, benzodiazepines, cannabinoids, etc.) at Screening or Day -1.
11. Subject unwilling to avoid consumption of coffee and caffeine containing beverages within 48 hours prior to Day -1 until discharge from the clinical site.
12. Subject unwilling to avoid use of alcohol or alcohol-containing foods, medications or beverages, within 48 hours prior to Day -1 until discharge from the clinical site.
13. Donation of blood (> 500 mL) or blood products within 2 months (56 days) prior to Day -1.
14. Use of over-the-counter (OTC) medications, prescription medications, or herbal remedies from 14 days or 5 time their half-lives whatever is more, prior to Day -1 and vitamin from 7 days prior to Day -1, until End-of-Study. By exception, acetaminophen 1000 mg per day is permitted.
15. Use of any drugs that induce or inhibit cytochrome P450 or P-glycoprotein within 30 days prior to dosing.
16. Any intake of grapefruit, grapefruit juice, Seville oranges, Seville orange marmalade, or other products containing grapefruit or Seville oranges within 7 days of dosing.
17. Use of an investigational drug within 30 days prior to Day 1.
18. Unwilling to abstain from vigorous exercise from 48 hours prior to Day -1 until End-of-Study.
19. Subject has a history of hypersensitivity to the investigational medicinal products (IMPs) or any of the excipients or to medicinal products with similar chemical structures.
20. Planning to father a child or donate sperm during the study and within 3 months following dosing.
21. Subject does not have veins suitable for cannulation or multiple venipunctures.
22. Subject is unable to understand the protocol requirements, instructions and study related restrictions, the nature, scope and possible consequences of the clinical study.
23. Subject is unlikely to comply with the protocol requirements, instructions and study related restrictions; e.g., uncooperative attitude, inability to return for Follow-up visits and improbability of completing the clinical study.
24. Subject has previously been enrolled in this clinical study.
25. Subjects involved in the planning or conduct of this clinical study.
26. Vulnerable subject (e.g. kept in detention)

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2013-08; Primary Completion 2014-03 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
The safety of GCC-4401C when repeatedly administered to healthy male adults | Up to 17 ~ 19 days after administration
  The following safety parameters will be recorded at regular intervals during the clinical study_
  * Vital signs (supine blood pressure (BP) and pulse, oral body temperature, respiratory rate (RR))
  * Twelve-lead ECG
  * 24-hour telemetry
  * Clinical laboratory testing (hematology, clinical chemistry, coagulation and urinalysis)
  * Hemoccult test
  * Adverse event assessments
  * Concomitant medication assessments
  * Physical examinations

SECONDARY OUTCOMES:
The Pharmacokinetics (PK) of GCC-4401C when repeatedly administered to healthy male adults | Predose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, and 48 hours post dose on Day 1 and Day 9 and at pre dose on Days 5 through 8
  The study consists of five cohorts (10 mg, 20 mg, 40 mg, 60 mg, and 80 mg) with eight subjects per cohort. In the 20 mg cohort, six additional subjects will receive rivaroxaban (Xarelto®) 20 mg as an active comparator in open-label fashion. Subjects will undergo dosing procedures on the morning of Day 1, and Day 3 to 9.
  * The following PK parameters for GCC-4401C and rivaroxaban will be determined after single dose, as appropriate_
    * Cmax
    * tmax
    * λz
    * Area under the curve from zero to the time of the last measurable concentration[AUC(0-last)]
    * Area under the curve from zero to infinity[AUC(0-inf)]
    * t½
    * Apparent systemic clearance(CL/F)
    * Vz/F
  * The following parameters will be determined after repeat treatment for the GCC-4401C and rivaroxaban_
    * Trough plasma concentration(Ctrough)
    * Cmax,ss,
    * Cmin,ss,
    * tmax,ss,
    * λz,ss,
    * AUC(0 τ),ss,
    * t½,ss,
    * CL

OTHER OUTCOMES:
The Pharmacodynamics (PD) of GCC-4401C when repeatedly administered to healthy male adults | predose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, and 48 hours post dose on Day 1 and Day 9
  The following PD parameters for GCC-4401C and rivaroxaban will be determined, as appropriate_
  * Activated partial thromboplastin time (aPTT)
  * Prothrombin time (PT)
  * International normalized ratio (INR)
  * Coagulation Factor X assay
  * Template bleeding time test
  * Low Molecular Weight Heparin (Factor Xa inhibition test)
  * Coagulation Factor X Chromogenic Activity Assay

CONTACTS AND LOCATIONS:
Overall Officials: David Han, M.D., Principal Investigator — California Clinical Trials Medical Group
Locations (1):
- PAREXEL Internatonal, Early Phase Clinical Unit _Los Angeles, California, United States